CLINICAL TRIAL: NCT01605071
Title: Time Past Menopause, Duration of Estrogen Deficiency, and Insulin Action
Brief Title: Timing Estrogen After MenoPaUSe
Acronym: TEMPUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 11-0788; R01DK088105 (NIH)
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Insulin Resistance
Keywords: menopause; estrogen; insulin sensitivity; estrogen receptors
MeSH Terms: conditions — Insulin Resistance | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Postmenopausal (Active Comparator): Postmenopausal women within 6 years of last menses who never used estrogen-based hormone therapy
  Interventions: Drug: Estradiol
- Late Postmenopausal (Active Comparator): Postmenopausal women more than 10 years since last menses who never used estrogen-based hormone therapy
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol — 1 week of transdermal estradiol (0.15mg)
  1 week of transdermal placebo
  Other Names: Climara

SUMMARY:
The aim of the current study is to test whether the effect of estrogen on insulin metabolism depends on the timing of treatment relative to when a woman went through menopause. The investigators hypothesize that estrogen will improve insulin sensitivity in early postmenopausal women, but decrease insulin sensitivity in late postmenopausal women.

DETAILED DESCRIPTION:
Large clinical trials have shown a reduced incidence of type 2 diabetes in postmenopausal women randomized to estrogen-based hormone therapy compared to placebo. Moreover, studies suggest development of diabetes is reduced in postmenopausal women who used hormone therapy for a part of the postmenopausal period compared to women who never used hormone therapy. Consistent with this, our preliminary data suggest that the timing of estrogen treatment relative to the menopause may be an important determinant of whether there are favorable effects on insulin action. Our observations suggest that estrogen improves insulin sensitivity in early postmenopausal women, but may decrease insulin sensitivity in those more than 10 years past menopause. More and more studies suggest estrogens have divergent effects on cardiovascular risk when initiated close to the onset of menopause rather than distant from the menopause; we hypothesize this is also true for diabetes risk. The goal of this study is to determine whether the effects of estrogen on insulin metabolism are different in women who are early postmenopausal compared to late postmenopausal. To meet our goal, we propose to measure insulin sensitivity in women who are within 6 years of the onset of menopause or more than 10 years beyond the menopause and who have not used hormone therapy previously. All women will be studied on two separate occasions, one day with and one day without short-term (1 week) treatment with transdermal estradiol. We expect that estradiol will increase insulin sensitivity in early postmenopausal women and decrease insulin sensitivity in late postmenopausal women. We also expect that estrogen receptors in fat and muscle may change with increasing time after menopause. Thus, we will collect fat and muscle biopsies to compare changes in estrogen receptors between early and late postmenopausal women and in response to 1 week of estradiol treatment. We believe these studies will provide evidence for a benefit of estradiol on insulin sensitivity when administered early, but not late, after menopause; likely contributing to delayed onset of type 2 diabetes in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* aged 45-70 yr
* postmenopausal (no menses ≥12 mo or bilateral oophorectomy and FSH >30 IU/L)
* ≤6yrs or ≥10yrs of menopause (last menses or oophorectomy)
* BMI <30 kg/m2 and weight stable (±2kg in past 2mo)
* non-smokers
* sedentary to moderately active (<3 days/wk of structured exercise)
* naïve to estrogen-based hormone therapies (previous use ≤6 months)
* CBC, CMP and TSH values within normal ranges specified by lab

Exclusion Criteria:

* underwent a partial hysterectomy (i.e., one or both ovaries left intact)
* underwent menopause (natural, chemical, or surgical) prior to age 45yr
* are between >6yr and <10yr of menopause (last menses or oophorectomy)
* previously used (>6 mo) or are currently using any formulation of estrogen-based HT (e.g., oral Premarin, transdermal 17beta-estradiol, selective estrogen receptor modulators)
* have T2DM or are being treated with glucose-lowering/ insulin sensitizing medications
* have uncontrolled hypertension (SBP>140 and/or DBP>90 mmHg)
* have hypertriglyceridemia (>400 mg/dL)
* have contraindications to estrogen therapy (history of venous thromboembolism, heart disease, myocardial infarction, hormone sensitive cancer)
* have contraindications to biopsies (severe anemia, blood clotting disorders)

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-09; Primary Completion 2015-11 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachael E Van Pelt, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Pelt RE, Schwartz RS, Kohrt WM. Insulin secretion and clearance after subacute estradiol administration in postmenopausal women. J Clin Endocrinol Metab. 2008 Feb;93(2):484-90. doi: 10.1210/jc.2007-1657. Epub 2007 Nov 6. PMID 17986638
- [Background] Kanaya AM, Herrington D, Vittinghoff E, Lin F, Grady D, Bittner V, Cauley JA, Barrett-Connor E; Heart and Estrogen/progestin Replacement Study. Glycemic effects of postmenopausal hormone therapy: the Heart and Estrogen/progestin Replacement Study. A randomized, double-blind, placebo-controlled trial. Ann Intern Med. 2003 Jan 7;138(1):1-9. doi: 10.7326/0003-4819-138-1-200301070-00005. PMID 12513038
- [Background] Bonds DE, Lasser N, Qi L, Brzyski R, Caan B, Heiss G, Limacher MC, Liu JH, Mason E, Oberman A, O'Sullivan MJ, Phillips LS, Prineas RJ, Tinker L. The effect of conjugated equine oestrogen on diabetes incidence: the Women's Health Initiative randomised trial. Diabetologia. 2006 Mar;49(3):459-68. doi: 10.1007/s00125-005-0096-0. Epub 2006 Jan 27. PMID 16440209
- [Background] Margolis KL, Bonds DE, Rodabough RJ, Tinker L, Phillips LS, Allen C, Bassford T, Burke G, Torrens J, Howard BV; Women's Health Initiative Investigators. Effect of oestrogen plus progestin on the incidence of diabetes in postmenopausal women: results from the Women's Health Initiative Hormone Trial. Diabetologia. 2004 Jul;47(7):1175-1187. doi: 10.1007/s00125-004-1448-x. Epub 2004 Jul 14. PMID 15252707
- [Background] Pentti K, Tuppurainen MT, Honkanen R, Sandini L, Kroger H, Alhava E, Saarikoski S. Hormone therapy protects from diabetes: the Kuopio osteoporosis risk factor and prevention study. Eur J Endocrinol. 2009 Jun;160(6):979-83. doi: 10.1530/EJE-09-0151. Epub 2009 Mar 25. PMID 19321660
- [Derived] Park YM, Keller AC, Runchey SS, Miller BF, Kohrt WM, Van Pelt RE, Kang C, Jankowski CM, Moreau KL. Acute estradiol treatment reduces skeletal muscle protein breakdown markers in early- but not late-postmenopausal women. Steroids. 2019 Jun;146:43-49. doi: 10.1016/j.steroids.2019.03.008. Epub 2019 Mar 27. PMID 30928279
- [Derived] Park YM, Pereira RI, Erickson CB, Swibas TA, Cox-York KA, Van Pelt RE. Estradiol-mediated improvements in adipose tissue insulin sensitivity are related to the balance of adipose tissue estrogen receptor alpha and beta in postmenopausal women. PLoS One. 2017 May 4;12(5):e0176446. doi: 10.1371/journal.pone.0176446. eCollection 2017. PMID 28472101
- [Derived] Pereira RI, Casey BA, Swibas TA, Erickson CB, Wolfe P, Van Pelt RE. Timing of Estradiol Treatment After Menopause May Determine Benefit or Harm to Insulin Action. J Clin Endocrinol Metab. 2015 Dec;100(12):4456-62. doi: 10.1210/jc.2015-3084. Epub 2015 Oct 1. PMID 26425886
- See also: IMAGE research group study website — http://medschool.ucdenver.edu/image

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Postmenopausal: Postmenopausal women within 6 years of last menses who never used estrogen-based hormone therapy
  Estradiol: 1 week of transdermal estradiol (0.15mg)
  1 week of transdermal placebo
- Late Postmenopausal: Postmenopausal women more than 10 years since last menses who never used estrogen-based hormone therapy
  Estradiol: 1 week of transdermal estradiol (0.15mg)
  1 week of transdermal placebo
Period: Overall Study
Arm/Group | Early Postmenopausal | Late Postmenopausal
Started (Includes those who were randomized and dropped or randomized, completed initial testing then dropped) | 27 | 26
Completed | 24 | 24
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Postmenopausal | Late Postmenopausal | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Customized [Count of Participants; unit: Participants]
  45-70 years of age | 22 | 24 | 46
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Insulin-mediated Glucose Disposal Rate (Hyperinsulinemic-euglycemic Clamp)
Description: Estrogen mediated change in glucose disposal rate and time since menopause
  * Baseline GDR (no difference between groups)
  * E2 mediated change (significant difference between groups)
  randomized order of testing, cross-over design
Time Frame: after 1wk estradiol or placebo
Measure: Mean (Standard Deviation); unit: mg/kg FFM/min
Arm/Group | Early Postmenopausal | Late Postmenopausal
Number analyzed (Participants) | 22 | 24
mg/kg FFM/min
  Placebo | 11.7 (2.8) | 11.5 (3.0)
  Estrogen | 12.2 (3.1) | 10.7 (2.9)

2. Secondary Outcome: Skeletal Muscle Estrogen Receptor Expression
Description: Estrogen receptors (ERα and ERβ) differences in time since menopause and estrogen treatment
  randomized order of testing, cross-over design
Time Frame: after 1wk estradiol or placebo
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Early Postmenopausal | Late Postmenopausal
Number analyzed (Participants) | 13 | 14
AU
  ERα nuclear protein (Placebo) | 1 (0.25) | 0.71 (0.20)
  ERα nuclear protein (Estrogen) | 0.92 (0.37) | 0.80 (0.31)
  ERβ nuclear protein (Placebo) | 1 (0.35) | 0.78 (0.26)
  ERβ nuclear protein (Estrogen) | 0.97 (0.47) | 0.75 (0.26)
  ERα cytosolic protein (Placebo) | 1 (0.40) | 1 (0.62)
  ERα cytosolic protein (Estrogen) | 0.63 (0.32) | 0.83 (0.45)
  ERβ cytosolic protein (Placebo) | 1 (0.41) | 0.7 (0.26)
  ERβ cytosolic protein (Estrogen) | 0.89 (0.44) | 0.64 (0.25)

3. Secondary Outcome: Skeletal Muscle Estrogen Receptor Expression (Protein/Cyto Protein)
Description: as for outcome 2
Time Frame: after 1wk estradiol or placebo
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Early Postmenopausal | Late Postmenopausal
Number analyzed (Participants) | 13 | 14
ratio
  ERα nuclear protein/cyto protein (Placebo) | 0.94 (0.34) | 0.78 (0.37)
  ERα nuclear protein/cyto protein (Estrogen) | 1.49 (0.92) | 0.98 (0.39)
  ERβ nuclear protein/cyto protein (Placebo) | 1 (0.53) | 1.13 (0.52)
  ERβ nuclear protein/cyto protein (Estrogen) | 1.13 (0.54) | 1.07 (0.39)

4. Secondary Outcome: Adipose Tissue Estrogen Receptor Expression
Description: Adipose tissue estrogen receptor expression associated with age and menopause
  Abdominal and femoral subcutaneous adipose tissue ERα and ERβ expression
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: 2ΔCT
Arm/Group | Early Postmenopausal | Late Postmenopausal
Number analyzed (Participants) | 23 | 22
2ΔCT
  Abdominal ERα (ESR1) | 1.58 (1.17) | 0.96 (0.58)
  Abdominal ERβ (ESR2) | 1.17 (0.70) | 1.22 (0.64)
  Femoral ERα (ESR1) | 1.44 (0.98) | 0.97 (0.49)
  Femoral ERβ (ESR2) | 1.09 (0.68) | 1.25 (0.71)

5. Secondary Outcome: Adipose Tissue Estrogen Receptor Expression (ERα:ERβ)
Description: Adipose tissue estrogen receptor expression associated with age and menopause
  Abdominal and femoral subcutaneous adipose tissue ratio of ERα:ERβ expression
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Early Postmenopausal | Late Postmenopausal
Number analyzed (Participants) | 23 | 22
ratio
  Abdominal ERα:ERβ (ESR1:ESR2) | 1.47 (0.71) | 0.89 (0.55)
  Femoral ERα:ERβ (ESR1:ESR2) | 1.143 (0.85) | 0.87 (0.37)

ADVERSE EVENTS:
Time Frame: 4 months participants were randomized in a crossover manner, visits were separated by approximately 2 months. - 1 week of placebo/study testing - 1 week of transdermal E2/study testing.
Description: No deaths or serious adverse events occurred in this study
Groups:
- Placebo: 1 week of transdermal placebo
- Estrogen: Estradiol: 1 week of transdermal estradiol (0.15mg)
Arm/Group | Placebo | Estrogen
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 6/37 | 2/37
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=37) | Estrogen (N=37)
Migraine/nausea (General disorders) | 2 (2) | 0 (0) — Migraine/nausea
bruising/discomfort (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Bruising/discomfort at biopsy site
CT scan abnormality (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Incidental finding at baseline, not related to the study
Irritation at IV site (General disorders) | 1 (1) | 0 (0)
Extended E2 administration (General disorders) | 0 (0) | 1 (1)
Low pulse (General disorders) | 1 (1) | 0 (0)
IV infiltration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No